CLINICAL TRIAL: NCT01200979
Title: Assessment of Alterations in Immune Function During Pregnancy and Post Parturition
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 100205; 10-I-0205
Record Dates: First submitted 2010-09-11; First posted 2010-09-14 (Estimated); Last update posted 2019-10-18 (Actual); Status verified 2019-10-11

CONDITIONS: Pregnancy Immune Function
Keywords: Gene Expression; IN VITRO; Immunosuppression; Infection; Neutrophils; Pregnancy; Immune Function
MeSH Terms: conditions — Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (2):
- pregnant flu vaccinated: pregnant women that choose to receive the seasonal flu vaccine
- pregnant non-flu vaccinated: pregnant women that do not receive the flu vaccine

SUMMARY:
Traditionally, it has been suggested that pregnancy causes an immunosuppressive state that would facilitate fetal tolerance and result in an increased susceptibility to infection. Although the suppression has been characterized as a global T-cell defect, the observation that the increase in susceptibility is restricted only to specific intracellular bacteria and viruses is consistent with a down regulation of only certain components of the innate immune system. Progress in the treatment and management of infections during pregnancy will require further understanding of the changes to the immune system that occur during pregnancy. It is hypothesized that there is a fundamental down-regulation in the innate immune system that occurs during pregnancy and remains until delivery and that changes in serum cytokines influence na(SqrRoot) ve CD4 differentiation to different subpopulations. To that end, this study will evaluate blood samples drawn from pregnant women during early, mid, and late pregnancy and post-partum for changes in the innate immune system and compare them to those of healthy, non-pregnant women. Changes in the cytokine profile and in the lymphocyte and natural killer (NK) cell populations will be identified. A comparison of any observed changes will be made with those previously reported for in vitro and in vivo studies.

DETAILED DESCRIPTION:
Traditionally, it has been suggested that pregnancy causes an immunosuppressive state that would facilitate fetal tolerance and result in an increased susceptibility to infection. Although the suppression has been characterized as a global T-cell defect, the observation that the increase in susceptibility is restricted only to specific intracellular bacteria and viruses is consistent with a down regulation of only certain components of the innate immune system. Progress in the treatment and management of infections during pregnancy will require further understanding of the changes to the immune system that occur during pregnancy. It is hypothesized that there is a fundamental down-regulation in the innate immune system that occurs during pregnancy and remains until delivery and that changes in serum cytokines influence na(SqrRoot) ve CD4 differentiation to different subpopulations. To that end, this study will evaluate blood samples drawn from pregnant women during early, mid, and late pregnancy and post-partum for changes in the innate immune system and compare them to data on a similar cohort of women of childbearing age from an existing database of healthy, non-pregnant women. Changes in the cytokine profile, gene expression by microarray, and in the lymphocyte and natural killer (NK) cell populations will be identified. We may perform neutrophil analysis. We will evaluate toll-like receptors functionality, and any changes in PBMC throughout pregnancy.

We also plan to evaluate serum cytokine panels, PBMC by flow cytometry, and PBMC for microarray of gene expression, before and after administration of the influenza vaccine in up to 20 of the 40 pregnant subjects. Antibody levels will be measured as well.

A comparison of any observed changes will be made with those previously reported for in vitro and in vivo studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

All pregnant study subjects must:

* Be between the ages of 18-45 years old.
* Have a positive pregnancy test (urine).
* Be of an estimated gestational age of between 10 and 20 weeks either by ultrasound or LMP.
* Have an identified primary care provider for the pregnancy.
* Be willing to sign the collaborative study consent form from CHI.
* Be willing to have samples collected and stored for future research and immunological studies
* Be willing to sign the collaborative study consent form for normal volunteers from CHI

Up to twenty pregnant subjects who agree to receive the seasonal influenza vaccine must:

* Have no history of allergic reaction to the vaccine or its contents
* Not have received the vaccine from other providers this flu season
* Agree to have an additional 20cc of blood drawn at both Day +1 and Day +7 post-vaccine for immune analysis.

EXCLUSION CRITIERIA:

A subject will be excluded if she:

* Has an identified underlying chronic medical condition that may adversely affect the immune system (e.g., autoimmune, HIV, or hematologic) or the need for immunomodulating medications (e.g., oral steroids) within 30 days prior to conception for a suspected immune disorder. Oral steroid use for any other reason must have been discontinued for at least 30 days prior to participation.
* Is found to have a Hemoglobin reading of less than 8g/dL.
* Has any other medical condition which, in the opinion of the Principal Investigator, poses an unacceptable risk to the subject s participation in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2011-09-30; Study Completion 2019-10-11

PRIMARY OUTCOMES:
Changes in lymphocyte and NK cell populations during pregnancy compared to non-pregnant control samples. | 1st, 2nd, and 3rd trimesters and postpartum and postpartum
  Changes in lymphocyte and NK cell populations during pregnancy compared to non- pregnant control samples. [Time Frame: 1st, 2nd, and 3rd trimesters and postpartum and postpartum]
Changes in Cytokine profiles during pregnancy | 1st, 2nd, and 3rd trimesters and postpartum and postpartum
  Changes in Cytokine profiles during pregnancy compared to non-pregnant control samples
Functionality of Toll-like receptors and changes in gene expression | 1st, 2nd, and 3rd trimesters and postpartum and postpartum
  Functionality of Toll-like receptors and changes in gene expression during pregnancy during pregnancy compared to non-pregnant control samples [Time Frame: 1st, 2nd, and 3rd trimesters and postpartum]

SECONDARY OUTCOMES:
Functionality of Toll-like receptors and changes in gene expression | Before and after the administration of the influenza vaccine in a subset of pregnant women
  Functionality of Toll-like receptors and changes in gene expression during pregnancy during pregnancy compared to non-pregnant control samples, in a subset of pregnant women [Time Frame: Before and after the administration of the influenza vaccine in a subset of pregnant women]
Changes in lymphocyte and INK cell populations | Before and after the administration of the influenza vaccine in a subset of pregnant women
  Changes in lymphocyte and INK cell populations during pregnancy compared to non-pregnant control samples, in a subset of pregnant women [Time Frame: Before and after the administration of the influenza vaccine in a subset of pregnant women]
Changes in Cytokine profiles | Before and after the administration of the influenza vaccine in a subset of pregnant women
  Changes in Cytokine profiles during pregnancy compared to non-pregnant control samples, in a subset of pregnant women [Time Frame: Before and after the administration of the influenza vaccine in a subset of pregnant women]

CONTACTS AND LOCATIONS:
Overall Officials: Christa S Zerbe, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Pejcic-Karapetrovic B, Gurnani K, Russell MS, Finlay BB, Sad S, Krishnan L. Pregnancy impairs the innate immune resistance to Salmonella typhimurium leading to rapid fatal infection. J Immunol. 2007 Nov 1;179(9):6088-96. doi: 10.4049/jimmunol.179.9.6088. PMID 17947683
- [Background] Luppi P. How immune mechanisms are affected by pregnancy. Vaccine. 2003 Jul 28;21(24):3352-7. doi: 10.1016/s0264-410x(03)00331-1. PMID 12850338
- [Background] Zhao J, Lei Z, Liu Y, Li B, Zhang L, Fang H, Song C, Wang X, Zhang GM, Feng ZH, Huang B. Human pregnancy up-regulates Tim-3 in innate immune cells for systemic immunity. J Immunol. 2009 May 15;182(10):6618-24. doi: 10.4049/jimmunol.0803876. PMID 19414817